CLINICAL TRIAL: NCT04752371
Title: A Phase 1b, Multicenter, Open-Label Study to Evaluate the Safety and Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Camoteskimab in Subjects With Adult Onset Still's Disease
Brief Title: A Study to Evaluate Camoteskimab in Participants With Still's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor discretion
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AEVI-007-AOSD-101; 2020-004099-16 (EudraCT Number)
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Adult Onset Still's Disease
Keywords: Adult Onset Still's Disease; AEVI-007; Camoteskimab; IL-18; sJIA
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Camoteskimab 7 mg/kg (Experimental): 6 participants will be administered camoteskimab at a dose of 7 mg/kg (500 mg maximum) at Baseline, Week 4, and Week 8.
  Interventions: Drug: Camoteskimab (CERC-007, AVTX-007, AEVI-007)
- Cohort 2: Camoteskimab Dose escalation/reduction (Experimental): Cohort 2 dose will be determined based on a review of Cohort 1 data. 6 participants will be administered camoteskimab at the determined dose at Baseline, Week 4, and Week 8.
  Interventions: Drug: Camoteskimab (CERC-007, AVTX-007, AEVI-007)

INTERVENTIONS:
Drug: Camoteskimab (CERC-007, AVTX-007, AEVI-007) — Intravenous (IV) Infusion

SUMMARY:
The main purpose of the study is to evaluate the safety and tolerability of Camoteskimab in participants with Still's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 75 years of age (inclusive) at the time of consent. The date of signature of the informed consent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the Screening Visit (Visit 1).
2. Subject has been diagnosed with AOSD based on classification criteria (according to Yamaguchi et al, 1992) defined as having 5 or more of the following criteria, 2 of which are major:

   a. Major Criteria i. Fever >39°C, lasting 1 week or longer ii. Arthralgia or arthritis, lasting 2 weeks or longer iii. Typical rash iv. Leukocytes >10,000 mm3 with >80% polymorphonuclear cells b. Minor Criteria i. Sore throat ii. Recent development of significant lymphadenopathy iii. Hepatomegaly or splenomegaly iv. Abnormal liver function tests v. Negative tests for antinuclear antibody and rheumatoid factor
3. Subject has reported a recurring fever >38°C, consistent with active disease, within the last 5 days of the Screening and Baseline Visits.
4. If undergoing treatment with non-steroidal anti-inflammatory drugs (NSAID), subject is on a stable dose for at least 48 hours prior to the Baseline Visit (Visit 2).
5. If undergoing treatment with glucocorticoids, subject is on a stable dose for at least 48 hours prior to the Baseline Visit (Visit 2).
6. If undergoing treatment with conventional disease-modifying anti-rheumatic drugs (DMARDs), subject is on a stable dose for at least 4 weeks prior to the Baseline Visit (Visit 2).
7. For subjects who have received treatment with biological DMARDs, subject has the required washout (normalization) period prior to the Baseline Visit (Visit 2).

   The washout (normalization) period for biological DMARDs is as follows:
   1. Anakinra - 1 week
   2. Etanercept, rilonacept - 4 weeks
   3. Adalimumab, certolizumab, infliximab, golimumab, abatacept, tocilizumab and canakinumab - 8 weeks
   4. Rituximab - 36 weeks
8. Non-pregnant female subjects of childbearing potential who are heterosexually active and non-sterile male subjects with female sexual partners of childbearing potential agree to use a highly effective method of contraception during treatment and for 25 weeks following the last dose of investigational product. A highly effective method of birth control is defined as one that results in a low failure rate (ie, <1% per year) when used consistently and correctly, such as oral/injectable/inserted/implanted/transdermal contraceptives, intrauterine hormone-releasing system or intrauterine device (IUD), or sexual abstinence. Contraception is not required where at least 6 weeks has passed since sterilization, defined as females having undergone one of the following surgeries: hysterectomy, bilateral tubal ligation or occlusion, bilateral oophorectomy, or bilateral salpingectomy; and males who are vasectomized. Contraception is also not required where females are postmenopausal (defined as 12 consecutive months of spontaneous amenorrhea and age ≥51 years). Females of reproductive potential must have a negative pregnancy test as part of the screening/baseline assessment.
9. Subject has provided written informed consent for this study.
10. Subject is willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is, in the opinion of the investigator, mentally or legally incapacitated, or has significant emotional problems at the time of the Screening Visit (Visit 1) that could interfere with the subject's participation or cooperation with the conduct of study evaluations
2. Subject has a chronic severe or uncontrolled medical disorder that might confound the results of safety assessments conducted in the study in the opinion of the Investigator or Medical Monitor.
3. Subject has another serious chronic-inflammatory disease.
4. Subject has a relevant, active infection or another disease, which entails a tendency towards infection.
5. Subject has active macrophage activation syndrome.
6. Subject has a history of unresolved latent tuberculosis.
7. Subject has the following abnormal values:

   1. Serum creatinine concentration >1.5 mg/dl.
   2. Hemoglobin ≤ 10 g/dl, neutrophils ≤1,500/μl and/or thrombocytes ≤75,000/μl.
8. Subject has a history of neoplasia with the exception of a curatively treated non-melanoma skin tumor or carcinoma of the cervix treated in situ without any indication of recurrence within the last 10 years.
9. Subject has received a vaccination with a live vaccine within 12 weeks prior to the Baseline Visit (Visit 2).
10. Subject has used an investigational product or been enrolled in a clinical study including vaccines within 30 days of the Screening Visit (Visit 1).
11. Subject has known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any ingredients of the investigational product.
12. Subject is pregnant or is breastfeeding and will not abstain from breastfeeding during participation in the study and for 25 weeks post last dose of investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs | Baseline to Week 24
Incidence of Clinically Significant Changes from Baseline in Vital Signs | Baseline to Week 24
Incidence of Clinically Significant Changes from Baseline in Clinical Laboratory Results | Baseline to Week 24

SECONDARY OUTCOMES:
Proportion of subjects who achieved absence of fever | Baseline to Week 24
  Fever defined as no temperature > 38 degrees Celcius for 48 hours
Proportion of subjects whose C-Reactive Protein (CRP) Levels Reduced by 50% or more from Baseline | Baseline to Week 4 and Week 12
Change from Baseline in the Physician Global Assessment of Disease Activity | Baseline to Week 4 and Week 12
  Physician global assessment of disease activity will be assessed using a Visual Analogue Scale (VAS) where 0 mm indicates no evidence of disease and 100 mm indicates very severe disease activity.
Change from Baseline in the Patient Global Assessment of Disease Activity | Baseline to Week 4 and Week 12
  Patient global assessment of disease activity will be assessed using a Visual Analogue Scale (VAS) where 0 mm indicates no evidence of disease and 100 mm indicates very severe disease activity.
Change from Baseline in the modified Pouchot score | Baseline to Week 4 and Week 12
Change from Baseline in the Disease Activity Score-28 with C-Reactive Protein (DAS28-CRP) | Baseline to Week 4 and Week 12
Change from Baseline in CRP, ferritin, and ESR | Baseline to Week 4 and Week 12
Serum Concentration of camoteskimab | Baseline through Week 24

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - Sponsor Investigative Site, Gainesville, Florida
  - Sponsor Investigative Site, Ann Arbor, Michigan
- Sponsor Investigative Site, Ghent, Oost-Vlaanderen, Belgium
- Poland (3):
  - Sponsor Investigative Site, Elblag
  - Sponsor Investigative Site, Pomorskie
  - Sponsor Investigative Site, Poznan
- Ukraine (4):
  - Sponsor Investigative Site, Kyiv
  - Sponsor Investigative Site, Poltava
  - Sponsor Investigative Site, Ternopil
  - Sponsor Investigative Site, Vinnitsa

IPD SHARING:
Plan to Share IPD: No